CLINICAL TRIAL: NCT02761837
Title: The Breathe Well Program to Improve Asthma Outcomes
Brief Title: The Breathe Well Program for Adults With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: National Jewish Health
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either 1) usual care or 2) Interactive Voice Response (IVR) or 3) email. Those in the groups 2 or 3 will receive the intervention only if they smoke, underuse controller medication, or overuse rescue medication.
Masking Description: This is a pragmatic controlled trial. Participants randomized to the intervention group will know when they receive the intervention, which will consist of an automated contact by IVR call/text, or email.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVR call/text (Active Comparator): Identify gaps in care and contact patients by IVR phone call or text
  Interventions: Behavioral: IVR call/text
- Email (Active Comparator): Identify gaps in care and contact patients by email
  Interventions: Behavioral: Email

INTERVENTIONS:
Behavioral: IVR call/text — For patients under filling their inhaled corticosteroid or overusing B-agonist, the patient is contacted via IVR call or text
  Arms: IVR call/text
Behavioral: Email — Patients under filling their inhaled corticosteroid or overusing B-agonist, the the patient is contacted via email
  Arms: Email

SUMMARY:
The Breathe Well Study is a pragmatic, controlled trial to assess the effectiveness, cost-effectiveness, and implementation of the Breathe Well intervention, which combines evidence-based EHR and interactive behavior-change technologies (IBCT) and team-based care to improve asthma outcomes.

DETAILED DESCRIPTION:
Breathe Well uses the Kaiser Permanente Electronic Health Record (EHR) to identify asthma exacerbation risk factors. For patients with a history of frequent exacerbations or B-agonist overuse, the EHR notifies a nurse who uses an EHR-generated tailored clinical report and patient directed decision support tool to engage and empower patients to develop an action plan in collaboration with providers. EHR-templated notes and order sets facilitate care plan execution. Poor controller medication adherence or unaddressed smoking results in the patient being automatically enrolled in an IBCT medication refill or smoking cessation program. Breathe Well uses multiple EHR functions and a patient and provider team to address barriers to evidence-based asthma care for providers.The study will be conducted in 26 primary care clinics of Kaiser Permanente Colorado (KPCO) using a pragmatic clinical trial design. Up to 15,000 high-risk asthma patients will be assigned to Breathe Well or guideline-based usual care based on their clinic.

ELIGIBILITY:
Inclusion Criteria: Adults with ≥1 EHR of these indicators of an asthma care gap in the EHR will be eligible.

1. B-agonist overfilling
2. inhaled corticosteroid (ICS) underfilling
3. current smoker
4. asthma exacerbation in the last year

Exclusion Criteria:

1. limited life expectancy
2. diagnosis of chronic obstructive pulmonary disease
3. lack of a pharmacy benefit because medication use cannot be captured.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14978 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Asthma Exacerbations | 12 months
  Defined as number of urgent care visits, hospitalizations, or prescriptions of an oral corticosteroid

SECONDARY OUTCOMES:
Controller medication adherence | 12 months
  Days of medication possession will be calculated for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente of Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bender BG, Cvietusa PJ, Goodrich GK, King DK, Shoup JA. Adapting adaptive design methods to accelerate adoption of a digital asthma management intervention. Transl Behav Med. 2023 Apr 3;13(3):149-155. doi: 10.1093/tbm/ibac093. PMID 36689336
- [Derived] Cvietusa PJ, Wagner NM, Shoup JA, Goodrich GK, Shetterly SM, King DK, Raebel MA, Riggs CS, Bender B. Digital Communication Technology: Does Offering a Choice of Modality Improve Medication Adherence and Outcomes in a Persistent Asthma Population? Perm J. 2020 Dec;25:1. doi: 10.7812/TPP/20.189. PMID 33635779